CLINICAL TRIAL: NCT06882642
Title: Sensory Integration Therapy in a Sample of Children With Autism Spectrum Disorder; an Outcome Study
Brief Title: Sensory Integration Therapy in a Sample of Children With Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rahaf Mohamed Abdelrahman, Assistant Lecturer of Neurology and Psychiatry, Faculty of Medicine, Ain Shams University, Cairo, Egypt., Ain Shams University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMASU MD71/2023
Record Dates: First submitted 2025-02-27; First posted 2025-03-18 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Autism Spectrum Disorder; Children; Therapy
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sensory integration therapy (Experimental): Autistic patients will undergo sensory integration therapy
  Interventions: Procedure: Sensory integration therapy

INTERVENTIONS:
Procedure: Sensory integration therapy — Autistic patients will undergo sensory integration therapy

SUMMARY:
The objective of this study is to determine the effects of therapy in sensory rooms with multisensory environment on the severity of autism spectrum disorder and stereotyped and repetitive behaviours in a sample of Egyptian children with autism spectrum disorder

DETAILED DESCRIPTION:
Autism Spectrum Disorder is a neurodevelopmental disorder characterized by deficits in social interactions, social communication and stereotyped behaviours associated with sensory disorders occurring before the age of 3.

According to DSM-5, sensory processing disorders include hyper-reactivity to sensory stimuli which is an adverse response to sensory stimuli (specific sounds or textures, excessive smells), hypo-reactivity as an apparent indifference to sensory stimuli (pain or temperature-hot/cold) and sensory seeking as a strong desire for sensory intake (touching of objects, visual fascination with lights and movements) or unusual sensory interests in the environment.] Multisensory interactions in spatial processing are investigated with functional neuroimaging and electrophysiological recordings. Using fMRI, researchers identified candidate multisensory areas by looking for regions of cortex that are activated by visual and tactile stimuli, showing that multisensory processing in the human brain involves the multisensory areas of ''association'' cortex as well as the modality-specific areas of cortex that are specialized for the processing of stimulus features such as colour, shape and texture.

Ayres Sensory Integration therapy (ASI) is an individualized intervention designed to address the specific underlying sensory-motor issues that may be affecting children's performance during daily routines and activities, including participation within the classroom and in other contexts of the school.

ELIGIBILITY:
Inclusion Criteria:

* All patients included in the study are diagnosed with Autism spectrum disorder according to DSM-V criteria.
* Participants have to have a sensory problem in their diagnostic criteria.
* Age ranges between 3-10 years. (as scope of the study is focused on children)
* Both males and females.
* Parents or guardian agreed to informed consent.

Exclusion Criteria:

* Parents refusing to participate in the research
* Children with comorbid psychiatric and/or neurological disorder
* Children with co-morbid sensory deficit, hearing , vision, and motor deficit
* Intelligence quotient level below 60
* Children who scored typical performance in the sensory profile care-giver questionnaire

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-03-28 (Actual)

PRIMARY OUTCOMES:
Effect of sensory integration therapy | 12 weeks
  Effect of sensory integration therapy on autism spectrum disorder symptoms and signs and severity. The sessions are held weekly for 12 weeks, lasting half an hour, and the measurement is done before and after them, taking an hour. The sensory integration program lasts 12 weeks with 12 sessions, each 30 minutes. Participants must attend at least 9 sessions. Afterward, they will be reassessed using CARS and the Sensory Profile Caregiver questionnaire. The sensory room provides multisensory stimulation through tools like projectors, fibre optics, and auditory devices.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author after the end of study for one year.